CLINICAL TRIAL: NCT00696241
Title: A Phase 3, Double-Blind, Randomized, Placebo-Controlled Study to Evaluate the Efficacy and Safety of TAK-491 in Subjects With Essential Hypertension
Brief Title: Efficacy and Safety of Azilsartan Medoxomil in Participants With Essential Hypertension
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Takeda (Industry)
Responsible Party: Sr. VP, Clinical Science, Takeda Global Research & Development Center, Inc.
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 01-05-TL-491-008; U1111-1113-8905 (Registry Identifier: WHO)
Record Dates: First submitted 2008-06-10; First posted 2008-06-12 (Estimated); Results first posted 2011-04-19 (Estimated); Last update posted 2011-07-29 (Estimated); Status verified 2011-07

CONDITIONS: Hypertension
Keywords: Essential Hypertension; Cardiovascular Disease; High Blood Pressure; Drug Therapy
MeSH Terms: conditions — Hypertension; Essential Hypertension; Cardiovascular Diseases | interventions — azilsartan medoxomil; olmesartan; azilsartan; Olmesartan Medoxomil

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (5):
- Azilsartan Medoxomil 20 mg QD (Experimental)
  Interventions: Drug: Azilsartan medoxomil and olmesartan
- Azilsartan Medoxomil 40 mg QD (Experimental)
  Interventions: Drug: Azilsartan medoxomil and olmesartan
- Azilsartan Medoxomil 80 mg QD (Experimental)
  Interventions: Drug: Azilsartan medoxomil and olmesartan
- Olmesartan 40 mg QD (Active Comparator)
  Interventions: Drug: Olmesartan
- Placebo QD (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Azilsartan medoxomil and olmesartan — Azilsartan medoxomil 20 mg, tablets, azilsartan medoxomil 40 mg placebo-matching tablets, azilsartan medoxomil 80 mg placebo-matching tablets and olmesartan 40 mg placebo-matching tablets, orally, for up to 6 weeks.
  Other Names: TAK-491; Edarbi
  Arms: Azilsartan Medoxomil 20 mg QD
Drug: Azilsartan medoxomil and olmesartan — Azilsartan medoxomil 40 mg, tablets, azilsartan medoxomil 20 mg placebo-matching tablets, azilsartan medoxomil 80 mg placebo-matching tablets and olmesartan 40 mg placebo-matching tablets, orally, for up to 6 weeks.
  Other Names: TAK-491; Edarbi
  Arms: Azilsartan Medoxomil 40 mg QD
Drug: Azilsartan medoxomil and olmesartan — Azilsartan medoxomil 80 mg, tablets, azilsartan medoxomil 20 mg placebo-matching tablets, azilsartan medoxomil 40 mg placebo-matching tablets and olmesartan 40 mg placebo-matching tablets, orally, once daily for up to 6 weeks.
  Other Names: TAK-491; Edarbi
  Arms: Azilsartan Medoxomil 80 mg QD
Drug: Olmesartan — Olmesartan 40 mg, tablets, azilsartan medoxomil 20 mg placebo-matching tablets, azilsartan medoxomil 40 mg placebo-matching tablets and azilsartan medoxomil 80 mg placebo-matching tablets, orally, once daily for up to 6 weeks.
  Other Names: Benicar®
  Arms: Olmesartan 40 mg QD
Drug: Placebo — Azilsartan medoxomil 20 mg placebo-matching tablets, azilsartan medoxomil 40 mg placebo-matching tablets, azilsartan medoxomil 80 mg placebo-matching tablets, and olmesartan 40 mg placebo- matching tablets, orally, once daily for up to 6 weeks.
  Arms: Placebo QD

SUMMARY:
The purpose of this study is to determine the safety and efficacy of azilsartan medoxomil, once daily (QD), compared to placebo and olmesartan in participants with essential hypertension.

DETAILED DESCRIPTION:
Hypertension affects approximately 50 million individuals in the United States. As the population ages, the prevalence of hypertension will continue to increase if broad and effective preventive measures are not implemented. According to the World Health Organization, hypertension is the most common attributable cause of preventable death in developed nations, as uncontrolled hypertension greatly increases the risk of cardiovascular disease, cerebrovascular disease, and renal failure. Despite the availability of antihypertensive treatments, hypertension remains inadequately controlled; only about one-third of patients continue to maintain control successfully.

TAK-491 (azilsartan medoxomil) is an angiotensin II receptor blocker and this study is being conducted to evaluate the efficacy and safety of oral azilsartan medoxomil compared to placebo and olmesartan in subjects with essential hypertension.

Individuals who want to participate in this study will be required to provide written informed consent. Study participation is anticipated to be about 11 weeks. Multiple procedures will occur at each visit which may include fasting, blood collection, urine collection, vital signs including sitting blood pressure and pulse, body height and weight, physical examinations and electrocardiograms. Outside of the study center, participants will be required to wear an ambulatory blood pressure monitoring device at 24 hour intervals.

ELIGIBILITY:
Inclusion Criteria

1. Has essential hypertension (defined as sitting trough clinic systolic blood pressure between 150 and 180 mm Hg, inclusive at Day minus 1) and 24-hour mean systolic blood pressure greater than or equal to 130 mm Hg and less than or equal to 170 mm Hg at Day 1).
2. Females of childbearing potential who are sexually active must agree to use adequate contraception, and can neither be pregnant nor lactating from Screening throughout the duration of the study.
3. Clinical laboratory evaluations (including clinical chemistry, hematology, and complete urinalysis) within the reference range for the testing laboratory or the results are deemed not clinically significant for inclusion into this study by the investigator.
4. The subject is willing to discontinue current antihypertensive medications at the Screening Day minus 21 visit. If the subject is on amlodipine prior to screening, the subject is willing to discontinue this medication at Screening Day minus 28.

Exclusion Criteria

1. Sitting trough clinic diastolic blood pressure greater than 114 mm Hg at Day minus 1.
2. Baseline 24-hour ambulatory blood pressure monitor reading of insufficient quality.
3. History of myocardial infarction, heart failure, unstable angina, coronary artery bypass graft, percutaneous coronary intervention, hypertensive encephalopathy, cerebrovascular accident, or transient ischemic attack.
4. Clinically significant cardiac conduction defects (eg, third degree atrioventricular block, left bundle branch block, sick sinus syndrome, atrial fibrillation or atrial flutter).
5. Hemodynamically significant left ventricular outflow obstruction due to aortic valvular disease.
6. Secondary hypertension of any etiology.
7. Is noncompliant (less than 70% or greater than 130%) with study medication during Placebo Run-In Period.
8. Severe renal dysfunction or disease (based on calculated creatinine clearance less than 30 mL/min/1.73 m2) at Screening.
9. Known or suspected unilateral or bilateral renal artery stenosis.
10. History of drug abuse (defined as illicit drug use) or a history of alcohol abuse (defined as regular or daily consumption of more than 2 alcoholic drinks per day) within the past 2 years.
11. History of cancer that has not been in remission for at least 5 years prior to the first dose of study drug. (This criterion does not apply to those subjects with basal cell or stage I squamous cell carcinoma of the skin).
12. Type 1 or poorly controlled type 2 diabetes mellitus (glycosylated hemoglobin greater than 8.0%) at Screening.
13. Alanine aminotransferase level greater than 2.5 times the upper limit of normal, active liver disease, or jaundice at Screening.
14. Hyperkalemia (defined as serum potassium greater than the upper limit of normal per the central laboratory) at Screening.
15. Upper arm circumference less than 24 cm or greater than 42 cm.
16. Works night (3rd) shift (defined as 11 PM to 7 AM).
17. Currently participating in another investigational study or has participated in an investigational study within 30 days prior to Screening.
18. Any other serious disease or condition at Screening (or Randomization) that would compromise subject safety, might affect life expectancy, or make it difficult to successfully manage and follow the subject according to the protocol.
19. Randomized in a previous azilsartan medoxomil study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1275 (Actual)
Dates: Start 2007-06; Primary Completion 2008-10 (Actual); Study Completion 2008-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: VP Clinical Science Strategy, Study Director — Takeda
Locations (85):
- United States (80):
  - Birmingham, Alabama
  - Huntsville, Alabama
  - Mesa, Arizona
  - Phoenix, Arizona
  - Tempe, Arizona
  - Little Rock, Arkansas
  - Tempe, Arkansas
  - Beverly Hills, California
  - Carmichael, California
  - Fountain Valley, California
  - Long Beach, California
  - Los Gatos, California
  - Orangevale, California
  - Sacramento, California
  - Santa Ana, California
  - Spring Valley, California
  - Tustin, California
  - Westlake Village, California
  - Colorado Springs, Colorado
  - Farmington, Connecticut
  - Hollywood, Florida
  - Jacksonville, Florida
  - Jupiter, Florida
  - Melbourne, Florida
  - Miami, Florida
  - Naples, Florida
  - Ocala, Florida
  - Pembroke Pines, Florida
  - Sarasota, Florida
  - St. Petersburg, Florida
  - Augusta, Georgia
  - Lawrenceville, Georgia
  - Chicago, Illinois
  - Melrose Park, Illinois
  - Naperville, Illinois
  - Round Lake Beach, Illinois
  - Valparaiso, Indiana
  - Wichita, Kansas
  - Erlanger, Kentucky
  - Lexington, Kentucky
  - Auburn, Maine
  - West Yarmouth, Massachusetts
  - Benzonia, Michigan
  - Chelsea, Michigan
  - Omaha, Nebraska
  - Trenton, New Jersey
  - Wildwood Crest, New Jersey
  - Albuquerque, New Mexico
  - Brooklyn, New York
  - Orangevale, New York
  - Rochester, New York
  - Burlington, North Carolina
  - Charlotte, North Carolina
  - Raleigh, North Carolina
  - Salisbury, North Carolina
  - Statesville, North Carolina
  - Wilmington, North Carolina
  - Winston-Salem, North Carolina
  - Kettering, Ohio
  - Lyndhurst, Ohio
  - Marion, Ohio
  - Norman, Oklahoma
  - Oklahoma City, Oklahoma
  - Altoona, Pennsylvania
  - Reading, Pennsylvania
  - Mt. Pleasant, South Carolina
  - Simpsonville, South Carolina
  - Taylors, South Carolina
  - Nashville, Tennessee
  - New Tazewell, Tennessee
  - Dallas, Texas
  - Houston, Texas
  - Lake Jackson, Texas
  - North Richland Hills, Texas
  - San Antonio, Texas
  - Draper, Utah
  - Burke, Virginia
  - Norfolk, Virginia
  - Tacoma, Washington
  - Madison, Wisconsin
- Argentina (2):
  - Provincia de Buenos Aires
  - Provincia de Cordoba
- Mexico (3):
  - Aguascalientes
  - Mexico City
  - San Luis Potosí City

REFERENCES:
- [Result] White WB, Weber MA, Sica D, Bakris GL, Perez A, Cao C, Kupfer S. Effects of the angiotensin receptor blocker azilsartan medoxomil versus olmesartan and valsartan on ambulatory and clinic blood pressure in patients with stages 1 and 2 hypertension. Hypertension. 2011 Mar;57(3):413-20. doi: 10.1161/HYPERTENSIONAHA.110.163402. Epub 2011 Jan 31. PMID 21282560
- [Result] Bakris GL, Sica D, Weber M, White WB, Roberts A, Perez A, Cao C, Kupfer S. The comparative effects of azilsartan medoxomil and olmesartan on ambulatory and clinic blood pressure. J Clin Hypertens (Greenwich). 2011 Feb;13(2):81-8. doi: 10.1111/j.1751-7176.2010.00425.x. PMID 21272195

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants enrolled at 147 investigative sites in Argentina, Mexico, Peru and the United States from 25 June 2007 to 08 October 2008.
Pre-assignment Details: Participants with essential hypertension were enrolled in one of five, once-daily (QD) treatment groups.
Groups:
- Azilsartan Medoxomil 20 mg QD: Azilsartan medoxomil 20 mg, tablets, orally, once daily for up to 6 weeks.
- Azilsartan Medoxomil 40 mg QD: Azilsartan medoxomil 40 mg, tablets, orally, once daily for up to 6 weeks.
- Azilsartan Medoxomil 80 mg QD: Azilsartan medoxomil 80 mg, tablets, orally, once daily for up to 6 weeks.
- Olmesartan 40 mg QD: Olmesartan 40 mg, tablets, orally, once daily for up to 6 weeks.
- Placebo QD: Placebo-matching tablets, orally, once daily for up to 6 weeks.
Period: Overall Study
Arm/Group | Azilsartan Medoxomil 20 mg QD | Azilsartan Medoxomil 40 mg QD | Azilsartan Medoxomil 80 mg QD | Olmesartan 40 mg QD | Placebo QD
Started | 283 | 283 | 285 | 282 | 142
Completed | 259 | 261 | 261 | 268 | 130
Not Completed | 24 | 22 | 24 | 14 | 12
Not completed — Adverse Event | 11 | 3 | 6 | 4 | 5
Not completed — Protocol Violation | 1 | 1 | 2 | 0 | 3
Not completed — Lost to Follow-up | 1 | 4 | 1 | 2 | 0
Not completed — Withdrawal by Subject | 4 | 8 | 6 | 1 | 0
Not completed — Lack of Efficacy | 1 | 5 | 4 | 5 | 3
Not completed — Other | 6 | 1 | 5 | 2 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Azilsartan Medoxomil 20 mg QD | Azilsartan Medoxomil 40 mg QD | Azilsartan Medoxomil 80 mg QD | Olmesartan 40 mg QD | Placebo QD | Total
Number analyzed (Participants) | 283 | 283 | 285 | 282 | 142 | 1275
Age Categorical [Number; unit: participants]
  <45 years | 32 | 29 | 37 | 32 | 11 | 141
  Between 45 and 64 years | 173 | 187 | 161 | 153 | 84 | 758
  ≥65 years | 78 | 67 | 87 | 97 | 47 | 376
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 150 | 141 | 136 | 142 | 66 | 635
  Male | 133 | 142 | 149 | 140 | 76 | 640

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in the 24-hour Mean Systolic Blood Pressure Measured by Ambulatory Blood Pressure Monitoring.
Description: The change in 24-hour mean systolic blood pressure measured at week 6 relative to baseline. Ambulatory blood pressure monitoring measures blood pressure at regular intervals throughout the day and night. The 24-hour mean is the average of all measurements recorded for 24 hours after dosing.
Time Frame: Baseline and Week 6.
Population: Full analysis set with last observation carried forward.
Measure: Least Squares Mean (Standard Error); unit: mmHg
Arm/Group | Azilsartan Medoxomil 20 mg QD | Azilsartan Medoxomil 40 mg QD | Azilsartan Medoxomil 80 mg QD | Olmesartan 40 mg QD | Placebo QD
Number analyzed (Participants) | 241 | 244 | 243 | 250 | 120
mmHg | -12.15 (0.709) | -13.48 (0.704) | -14.62 (0.706) | -12.56 (0.696) | -1.40 (1.004)
Statistical Analysis 1: Comparison: Azilsartan Medoxomil 20 mg QD vs Placebo QD; Test type: Superiority or Other; p < 0.001, ANCOVA — Postbaseline P-value was from ANCOVA with terms for treatment (as a factor) and baseline value (as a covariate). Unadjusted p-value presented. Overall 0.05 level of significance for multiple comparisons controlled using stepwise testing procedure; Mean Difference (Final Values) = -10.75, 95% CI [-13.17 to -8.34]
Statistical Analysis 2: Comparison: Azilsartan Medoxomil 40 mg QD vs Placebo QD; Test type: Superiority or Other; p < 0.001, ANCOVA — [p-value comment as in outcome 1, analysis 1]; Mean Difference (Final Values) = -12.08, 95% CI 2-sided [-14.48 to -9.67]
Statistical Analysis 3: Comparison: Azilsartan Medoxomil 80 mg QD vs Placebo QD; Test type: Superiority or Other; p < 0.001, ANCOVA — [p-value comment as in outcome 1, analysis 1]; Mean Difference (Final Values) = -13.21, 95% CI 2-sided [-15.62 to -10.81]
Statistical Analysis 4: Comparison: Azilsartan Medoxomil 20 mg QD vs Olmesartan 40 mg QD; Test type: Superiority or Other; p = 0.687, ANCOVA — [p-value comment as in outcome 1, analysis 1]; Mean Difference (Final Values) = 0.40, 95% CI 2-sided [-1.55 to 2.35]
Statistical Analysis 5: Comparison: Azilsartan Medoxomil 40 mg QD vs Olmesartan 40 mg QD; Test type: Superiority or Other; p = 0.352, ANCOVA — [p-value comment as in outcome 1, analysis 1]; Mean Difference (Final Values) = -0.92, 95% CI 2-sided [-2.87 to 1.02]
Statistical Analysis 6: Comparison: Azilsartan Medoxomil 80 mg QD vs Olmesartan 40 mg QD; Test type: Superiority or Other; p = 0.038, ANCOVA — [p-value comment as in outcome 1, analysis 1]; Mean Difference (Final Values) = -2.06, 95% CI 2-sided [-4.00 to -0.12]

2. Secondary Outcome: Change From Baseline in Mean Trough Clinic Sitting Systolic Blood Pressure
Description: The change in mean trough clinic sitting systolic blood pressure measured at final visit or week 6 relative to baseline.
Time Frame: Baseline and Week 6.
Population: Full analysis set with last observation carried forward.
Measure: Least Squares Mean (Standard Error); unit: mmHg
Arm/Group | Azilsartan Medoxomil 20 mg QD | Azilsartan Medoxomil 40 mg QD | Azilsartan Medoxomil 80 mg QD | Olmesartan 40 mg QD | Placebo QD
Number analyzed (Participants) | 274 | 276 | 279 | 280 | 140
mmHg | -14.28 (0.956) | -14.47 (0.952) | -17.58 (0.947) | -14.87 (0.945) | -2.06 (1.337)
Statistical Analysis 1: Comparison: Azilsartan Medoxomil 20 mg QD vs Placebo QD; Test type: Superiority or Other; p < 0.001, ANCOVA — [p-value comment as in outcome 1, analysis 1]; Mean Difference (Final Values) = -12.23, 95% CI 2-sided [-15.45 to -9.00]
Statistical Analysis 2: Comparison: Azilsartan Medoxomil 40 mg QD vs Placebo QD; Test type: Superiority or Other; p < 0.001, ANCOVA — [p-value comment as in outcome 1, analysis 1]; Mean Difference (Final Values) = -12.42, 95% CI 2-sided [-15.64 to -9.20]
Statistical Analysis 3: Comparison: Azilsartan Medoxomil 80 mg QD vs Placebo QD; Test type: Superiority or Other; p < 0.001, ANCOVA — [p-value comment as in outcome 1, analysis 1]; Mean Difference (Final Values) = -15.53, 95% CI 2-sided [-18.74 to -12.31]
Statistical Analysis 4: Comparison: Azilsartan Medoxomil 20 mg QD vs Olmesartan 40 mg QD; Test type: Superiority or Other; p = 0.662, ANCOVA — [p-value comment as in outcome 1, analysis 1]; Mean Difference (Final Values) = 0.59, 95% CI 2-sided [-2.05 to 3.22]
Statistical Analysis 5: Comparison: Azilsartan Medoxomil 40 mg QD vs Olmesartan 40 mg QD; Test type: Superiority or Other; p = 0.768, ANCOVA — [p-value comment as in outcome 1, analysis 1]; Mean Difference (Final Values) = 0.40, 95% CI 2-sided [-2.24 to 3.03]
Statistical Analysis 6: Comparison: Azilsartan Medoxomil 80 mg QD vs Olmesartan 40 mg QD; Test type: Superiority or Other; p = 0.043, ANCOVA — [p-value comment as in outcome 1, analysis 1]; Mean Difference (Final Values) = -2.71, 95% CI 2-sided [-5.34 to -0.09]

3. Secondary Outcome: Change From Baseline in the 24-hour Mean Diastolic Blood Pressure Measured by Ambulatory Blood Pressure Monitoring.
Description: The change in 24-hour mean diastolic blood pressure measured at week 6 relative to baseline. Ambulatory blood pressure monitoring measures blood pressure at regular intervals throughout the day and night. The 24-hour mean is the average of all measurements recorded for 24 hours after dosing.
Time Frame: Baseline and Week 6.
Population: Full analysis set with last observation carried forward.
Measure: Least Squares Mean (Standard Error); unit: mmHg
Arm/Group | Azilsartan Medoxomil 20 mg QD | Azilsartan Medoxomil 40 mg QD | Azilsartan Medoxomil 80 mg QD | Olmesartan 40 mg QD | Placebo QD
Number analyzed (Participants) | 241 | 244 | 243 | 250 | 120
mmHg | -7.47 (0.458) | -8.38 (0.455) | -8.61 (0.456) | -7.74 (0.449) | -0.69 (0.649)
Statistical Analysis 1: Comparison: Azilsartan Medoxomil 20 mg QD vs Placebo QD; Test type: Superiority or Other; p < 0.001, ANCOVA — P-value was from ANCOVA with terms for treatment (as a factor) and baseline value (as a covariate). Unadjusted p-value is presented; Mean Difference (Final Values) = -6.78, 95% CI 2-sided [-8.34 to -5.22]
Statistical Analysis 2: Comparison: Azilsartan Medoxomil 40 mg QD vs Placebo QD; Test type: Superiority or Other; p < 0.001, ANCOVA — [p-value comment as in outcome 3, analysis 1]; Mean Difference (Final Values) = -7.68, 95% CI 2-sided [-9.24 to -6.13]
Statistical Analysis 3: Comparison: Azilsartan Medoxomil 80 mg QD vs Placebo QD; Test type: Superiority or Other; p < 0.001, ANCOVA — [p-value comment as in outcome 3, analysis 1]; Mean Difference (Final Values) = -7.92, 95% CI 2-sided [-9.47 to -6.36]
Statistical Analysis 4: Comparison: Azilsartan Medoxomil 20 mg QD vs Olmesartan 40 mg QD; Test type: Superiority or Other; p = 0.679, ANCOVA — [p-value comment as in outcome 3, analysis 1]; Mean Difference (Final Values) = 0.27, 95% CI 2-sided [-0.99 to 1.52]
Statistical Analysis 5: Comparison: Azilsartan Medoxomil 40 mg QD vs Olmesartan 40 mg QD; Test type: Superiority or Other; p = 0.319, ANCOVA — [p-value comment as in outcome 3, analysis 1]; Mean Difference (Final Values) = -0.64, 95% CI 2-sided [-1.89 to 0.62]
Statistical Analysis 6: Comparison: Azilsartan Medoxomil 80 mg QD vs Olmesartan 40 mg QD; Test type: Superiority or Other; p = 0.172, ANCOVA — [p-value comment as in outcome 3, analysis 1]; Mean Difference (Final Values) = -0.87, 95% CI 2-sided [-2.13 to 0.38]

4. Secondary Outcome: Change From Baseline in Mean Trough Clinic Sitting Diastolic Blood Pressure
Description: The change in mean trough clinic sitting diastolic blood pressure measured at final visit or week 6 relative to baseline.
Time Frame: Baseline and Week 6.
Population: Full analysis set with last observation carried forward.
Measure: Least Squares Mean (Standard Error); unit: mmHg
Arm/Group | Azilsartan Medoxomil 20 mg QD | Azilsartan Medoxomil 40 mg QD | Azilsartan Medoxomil 80 mg QD | Olmesartan 40 mg QD | Placebo QD
Number analyzed (Participants) | 274 | 276 | 279 | 280 | 140
mmHg | -6.82 (0.535) | -6.86 (0.533) | -8.42 (0.530) | -6.91 (0.529) | 0.21 (0.749)
Statistical Analysis 1: Comparison: Azilsartan Medoxomil 20 mg QD vs Placebo QD; Test type: Superiority or Other; p < 0.001, ANCOVA — [p-value comment as in outcome 3, analysis 1]; Mean Difference (Final Values) = -7.02, 95% CI 2-sided [-8.83 to -5.22]
Statistical Analysis 2: Comparison: Azilsartan Medoxomil 40 mg QD vs Placebo QD; Test type: Superiority or Other; p < 0.001, ANCOVA — [p-value comment as in outcome 3, analysis 1]; Mean Difference (Final Values) = -7.07, 95% CI 2-sided [-8.87 to -5.27]
Statistical Analysis 3: Comparison: Azilsartan Medoxomil 80 mg QD vs Placebo QD; Test type: Superiority or Other; p < 0.001, ANCOVA — [p-value comment as in outcome 3, analysis 1]; Mean Difference (Final Values) = -8.62, 95% CI 2-sided [-10.42 to -6.82]
Statistical Analysis 4: Comparison: Azilsartan Medoxomil 20 mg QD vs Olmesartan 40 mg QD; Test type: Superiority or Other; p = 0.908, ANCOVA — [p-value comment as in outcome 3, analysis 1]; Mean Difference (Final Values) = 0.09, 95% CI 2-sided [-1.39 to 1.56]
Statistical Analysis 5: Comparison: Azilsartan Medoxomil 40 mg QD vs Olmesartan 40 mg QD; Test type: Superiority or Other; p = 0.956, ANCOVA — [p-value comment as in outcome 3, analysis 1]; Mean Difference (Final Values) = 0.04, 95% CI 2-sided [-1.43 to 1.52]
Statistical Analysis 6: Comparison: Azilsartan Medoxomil 80 mg QD vs Olmesartan 40 mg QD; Test type: Superiority or Other; p = 0.044, ANCOVA — [p-value comment as in outcome 3, analysis 1]; Mean Difference (Final Values) = -1.51, 95% CI 2-sided [-2.98 to -0.04]

5. Secondary Outcome: Change From Baseline in Daytime (6am to 10 pm) Mean Systolic Blood Pressure Measured by Ambulatory Blood Pressure Monitoring.
Description: The change in daytime (6am to 10pm) mean systolic blood pressure measured at week 6 relative to baseline. Ambulatory blood pressure monitoring measures blood pressure at regular intervals throughout the day and night. Daytime mean is the average of all measurements recorded between the hours of 6 am and 10 pm.
Time Frame: Baseline and Week 6.
Population: Full analysis set with last observation carried forward.
Measure: Least Squares Mean (Standard Error); unit: mmHg
Arm/Group | Azilsartan Medoxomil 20 mg QD | Azilsartan Medoxomil 40 mg QD | Azilsartan Medoxomil 80 mg QD | Olmesartan 40 mg QD | Placebo QD
Number analyzed (Participants) | 241 | 244 | 243 | 250 | 120
mmHg | -12.57 (0.751) | -13.75 (0.746) | -14.96 (0.747) | -12.73 (0.737) | -1.54 (1.064)
Statistical Analysis 1: Comparison: Azilsartan Medoxomil 20 mg QD vs Placebo QD; Test type: Superiority or Other; p < 0.001, ANCOVA — [p-value comment as in outcome 3, analysis 1]; Mean Difference (Final Values) = -11.03, 95% CI 2-sided [-13.59 to -8.48]
Statistical Analysis 2: Comparison: Azilsartan Medoxomil 40 mg QD vs Placebo QD; Test type: Superiority or Other; p < 0.001, ANCOVA — [p-value comment as in outcome 3, analysis 1]; Mean Difference (Final Values) = -12.20, 95% CI 2-sided [-14.75 to -9.65]
Statistical Analysis 3: Comparison: Azilsartan Medoxomil 80 mg QD vs Placebo QD; Test type: Superiority or Other; p < 0.001, ANCOVA — [p-value comment as in outcome 3, analysis 1]; Mean Difference (Final Values) = -13.41, 95% CI 2-sided [-15.97 to -10.86]
Statistical Analysis 4: Comparison: Azilsartan Medoxomil 20 mg QD vs Olmesartan 40 mg QD; Test type: Superiority or Other; p = 0.879, ANCOVA — [p-value comment as in outcome 3, analysis 1]; Mean Difference (Final Values) = 0.16, 95% CI 2-sided [-1.90 to 2.22]
Statistical Analysis 5: Comparison: Azilsartan Medoxomil 40 mg QD vs Olmesartan 40 mg QD; Test type: Superiority or Other; p = 0.334, ANCOVA — [p-value comment as in outcome 3, analysis 1]; Mean Difference (Final Values) = -1.01, 95% CI 2-sided [-3.07 to 1.04]
Statistical Analysis 6: Comparison: Azilsartan Medoxomil 80 mg QD vs Olmesartan 40 mg QD; Test type: Superiority or Other; p = 0.034, ANCOVA — [p-value comment as in outcome 3, analysis 1]; Mean Difference (Final Values) = -2.22, 95% CI 2-sided [-4.28 to -0.16]

6. Secondary Outcome: Change From Baseline in Daytime (6am to 10 pm) Mean Diastolic Blood Pressure Measured by Ambulatory Blood Pressure Monitoring.
Description: The change in daytime (6am to 10pm) mean diastolic blood pressure measured at week 6 relative to baseline. Ambulatory blood pressure monitoring measures blood pressure at regular intervals throughout the day and night. Daytime mean is the average of all measurements recorded between the hours of 6 am and 10 pm.
Time Frame: Baseline and Week 6.
Population: Full analysis set with last observation carried forward.
Measure: Least Squares Mean (Standard Error); unit: mmHg
Arm/Group | Azilsartan Medoxomil 20 mg QD | Azilsartan Medoxomil 40 mg QD | Azilsartan Medoxomil 80 mg QD | Olmesartan 40 mg QD | Placebo QD
Number analyzed (Participants) | 241 | 244 | 243 | 250 | 120
mmHg | -7.71 (0.490) | -8.43 (0.487) | -8.87 (0.488) | -7.82 (0.481) | -0.59 (0.695)
Statistical Analysis 1: Comparison: Azilsartan Medoxomil 20 mg QD vs Placebo QD; Test type: Superiority or Other; p < 0.001, ANCOVA — [p-value comment as in outcome 3, analysis 1]; Mean Difference (Final Values) = -7.12, 95% CI 2-sided [-8.79 to -5.45]
Statistical Analysis 2: Comparison: Azilsartan Medoxomil 40 mg QD vs Placebo QD; Test type: Superiority or Other; p < 0.001, ANCOVA — [p-value comment as in outcome 3, analysis 1]; Mean Difference (Final Values) = -7.84, 95% CI 2-sided [-9.51 to -6.18]
Statistical Analysis 3: Comparison: Azilsartan Medoxomil 80 mg QD vs Placebo QD; Test type: Superiority or Other; p < 0.001, ANCOVA — [p-value comment as in outcome 3, analysis 1]; Mean Difference (Final Values) = -8.28, 95% CI 2-sided [-9.94 to -6.61]
Statistical Analysis 4: Comparison: Azilsartan Medoxomil 20 mg QD vs Olmesartan 40 mg QD; Test type: Superiority or Other; p = 0.877, ANCOVA — [p-value comment as in outcome 3, analysis 1]; Mean Difference (Final Values) = 0.11, 95% CI 2-sided [-1.24 to 1.45]
Statistical Analysis 5: Comparison: Azilsartan Medoxomil 40 mg QD vs Olmesartan 40 mg QD; Test type: Superiority or Other; p = 0.369, ANCOVA — [p-value comment as in outcome 3, analysis 1]; Mean Difference (Final Values) = -0.62, 95% CI 2-sided [-1.96 to 0.73]
Statistical Analysis 6: Comparison: Azilsartan Medoxomil 80 mg QD vs Olmesartan 40 mg QD; Test type: Superiority or Other; p = 0.126, ANCOVA — [p-value comment as in outcome 3, analysis 1]; Mean Difference (Final Values) = -1.05, 95% CI 2-sided [-2.39 to 0.30]

7. Secondary Outcome: Change From Baseline in the Nighttime (12 am to 6 am) Mean Systolic Blood Pressure Measured by Ambulatory Blood Pressure Monitoring.
Description: The change in nighttime (12am to 6am) mean systolic blood pressure measured at week 6 relative to baseline. Ambulatory blood pressure monitoring measures blood pressure at regular intervals throughout the day and night. Nighttime mean is the average of all measurements recorded between the hours of 12 am and 6 am.
Time Frame: Baseline and Week 6.
Population: Full analysis set with last observation carried forward.
Measure: Least Squares Mean (Standard Error); unit: mmHg
Arm/Group | Azilsartan Medoxomil 20 mg QD | Azilsartan Medoxomil 40 mg QD | Azilsartan Medoxomil 80 mg QD | Olmesartan 40 mg QD | Placebo QD
Number analyzed (Participants) | 241 | 244 | 243 | 250 | 120
mmHg | -11.10 (0.781) | -12.39 (0.775) | -13.35 (0.777) | -12.13 (0.766) | -0.97 (1.105)
Statistical Analysis 1: Comparison: Azilsartan Medoxomil 20 mg QD vs Placebo QD; Test type: Superiority or Other; p < 0.001, ANCOVA — [p-value comment as in outcome 3, analysis 1]; Mean Difference (Final Values) = -10.13, 95% CI 2-sided [-12.79 to -7.48]
Statistical Analysis 2: Comparison: Azilsartan Medoxomil 40 mg QD vs Placebo QD; Test type: Superiority or Other; p < 0.001, ANCOVA — [p-value comment as in outcome 3, analysis 1]; Mean Difference (Final Values) = -11.43, 95% CI 2-sided [-14.07 to -8.78]
Statistical Analysis 3: Comparison: Azilsartan Medoxomil 80 mg QD vs Placebo QD; Test type: Superiority or Other; p < 0.001, ANCOVA — [p-value comment as in outcome 3, analysis 1]; Mean Difference (Final Values) = -12.38, 95% CI 2-sided [-15.03 to -9.73]
Statistical Analysis 4: Comparison: Azilsartan Medoxomil 20 mg QD vs Olmesartan 40 mg QD; Test type: Superiority or Other; p = 0.346, ANCOVA — [p-value comment as in outcome 3, analysis 1]; Mean Difference (Final Values) = 1.03, 95% CI 2-sided [-1.12 to 3.18]
Statistical Analysis 5: Comparison: Azilsartan Medoxomil 40 mg QD vs Olmesartan 40 mg QD; Test type: Superiority or Other; p = 0.811, ANCOVA — [p-value comment as in outcome 3, analysis 1]; Mean Difference (Final Values) = -0.26, 95% CI 2-sided [-2.40 to 1.88]
Statistical Analysis 6: Comparison: Azilsartan Medoxomil 80 mg QD vs Olmesartan 40 mg QD; Test type: Superiority or Other; p = 0.267, ANCOVA — [p-value comment as in outcome 3, analysis 1]; Mean Difference (Final Values) = -1.21, 95% CI 2-sided [-3.35 to 0.93]

8. Secondary Outcome: Change From Baseline in the Nighttime (12 am to 6 am) Mean Diastolic Blood Pressure Measured by Ambulatory Blood Pressure Monitoring.
Description: The change in nighttime (12am to 6am) mean diastolic blood pressure measured at week 6 relative to baseline. Ambulatory blood pressure monitoring measures blood pressure at regular intervals throughout the day and night. Nighttime mean is the average of all measurements recorded between the hours of 12 am and 6 am.
Time Frame: Baseline and Week 6.
Population: Full analysis set with last observation carried forward.
Measure: Least Squares Mean (Standard Error); unit: mmHg
Arm/Group | Azilsartan Medoxomil 20 mg QD | Azilsartan Medoxomil 40 mg QD | Azilsartan Medoxomil 80 mg QD | Olmesartan 40 mg QD | Placebo QD
Number analyzed (Participants) | 241 | 244 | 243 | 250 | 120
mmHg | -6.98 (0.533) | -7.90 (0.530) | -7.79 (0.531) | -7.62 (0.523) | -0.96 (0.755)
Statistical Analysis 1: Comparison: Azilsartan Medoxomil 20 mg QD vs Placebo QD; Test type: Superiority or Other; p < 0.001, ANCOVA — [p-value comment as in outcome 3, analysis 1]; Mean Difference (Final Values) = -6.03, 95% CI 2-sided [-7.84 to -4.21]
Statistical Analysis 2: Comparison: Azilsartan Medoxomil 40 mg QD vs Placebo QD; Test type: Superiority or Other; p < 0.001, ANCOVA — [p-value comment as in outcome 3, analysis 1]; Mean Difference (Final Values) = -6.94, 95% CI 2-sided [-8.75 to -5.13]
Statistical Analysis 3: Comparison: Azilsartan Medoxomil 80 mg QD vs Placebo QD; Test type: Superiority or Other; p < 0.001, ANCOVA — [p-value comment as in outcome 3, analysis 1]; Mean Difference (Final Values) = -6.84, 95% CI 2-sided [-8.65 to -5.03]
Statistical Analysis 4: Comparison: Azilsartan Medoxomil 20 mg QD vs Olmesartan 40 mg QD; Test type: Superiority or Other; p = 0.394, ANCOVA — [p-value comment as in outcome 3, analysis 1]; Mean Difference (Final Values) = 0.64, 95% CI 2-sided [-0.83 to 2.10]
Statistical Analysis 5: Comparison: Azilsartan Medoxomil 40 mg QD vs Olmesartan 40 mg QD; Test type: Superiority or Other; p = 0.712, ANCOVA — [p-value comment as in outcome 3, analysis 1]; Mean Difference (Final Values) = -0.27, 95% CI 2-sided [-1.74 to 1.19]
Statistical Analysis 6: Comparison: Azilsartan Medoxomil 80 mg QD vs Olmesartan 40 mg QD; Test type: Superiority or Other; p = 0.818, ANCOVA — [p-value comment as in outcome 3, analysis 1]; Mean Difference (Final Values) = -0.17, 95% CI 2-sided [-1.63 to 1.29]

9. Secondary Outcome: Change From Baseline in the 12-hour Mean Systolic Blood Pressure Measured by Ambulatory Blood Pressure Monitoring
Description: The change in the 12-hour mean systolic blood pressure measured at week 6 relative to baseline. Ambulatory blood pressure monitoring measures blood pressure at regular intervals throughout the day and night. The 12-hour mean is the average of all measurements recorded in the first 12 hours after dosing.
Time Frame: Baseline and Week 6.
Population: Full analysis set with last observation carried forward.
Measure: Least Squares Mean (Standard Error); unit: mmHg
Arm/Group | Azilsartan Medoxomil 20 mg QD | Azilsartan Medoxomil 40 mg QD | Azilsartan Medoxomil 80 mg QD | Olmesartan 40 mg QD | Placebo QD
Number analyzed (Participants) | 241 | 244 | 243 | 250 | 120
mmHg | -12.72 (0.795) | -14.05 (0.790) | -15.18 (0.791) | -13.07 (0.780) | -1.36 (1.126)
Statistical Analysis 1: Comparison: Azilsartan Medoxomil 20 mg QD vs Placebo QD; Test type: Superiority or Other; p < 0.001, ANCOVA — [p-value comment as in outcome 3, analysis 1]; Mean Difference (Final Values) = -11.35, 95% CI 2-sided [-14.05 to -8.64]
Statistical Analysis 2: Comparison: Azilsartan Medoxomil 40 mg QD vs Placebo QD; Test type: Superiority or Other; p < 0.001, ANCOVA — [p-value comment as in outcome 3, analysis 1]; Mean Difference (Final Values) = -12.68, 95% CI 2-sided [-15.38 to -9.98]
Statistical Analysis 3: Comparison: Azilsartan Medoxomil 80 mg QD vs Placebo QD; Test type: Superiority or Other; p < 0.001, ANCOVA — [p-value comment as in outcome 3, analysis 1]; Mean Difference (Final Values) = -13.81, 95% CI 2-sided [-16.51 to -11.11]
Statistical Analysis 4: Comparison: Azilsartan Medoxomil 20 mg QD vs Olmesartan 40 mg QD; Test type: Superiority or Other; p = 0.750, ANCOVA — [p-value comment as in outcome 3, analysis 1]; Mean Difference (Final Values) = 0.35, 95% CI 2-sided [-1.83 to 2.54]
Statistical Analysis 5: Comparison: Azilsartan Medoxomil 40 mg QD vs Olmesartan 40 mg QD; Test type: Superiority or Other; p = 0.378, ANCOVA — [p-value comment as in outcome 3, analysis 1]; Mean Difference (Final Values) = -0.98, 95% CI 2-sided [-3.16 to 1.20]
Statistical Analysis 6: Comparison: Azilsartan Medoxomil 80 mg QD vs Olmesartan 40 mg QD; Test type: Superiority or Other; p = 0.059, ANCOVA — [p-value comment as in outcome 3, analysis 1]; Mean Difference (Final Values) = -2.10, 95% CI 2-sided [-4.28 to 0.08]

10. Secondary Outcome: Change From Baseline in the 12-hour Mean Diastolic Blood Pressure Measured by Ambulatory Blood Pressure Monitoring
Description: The change in the 12-hour mean diastolic blood pressure measured at week 6 relative to baseline. Ambulatory blood pressure monitoring measures blood pressure at regular intervals throughout the day and night. The 12-hour mean is the average of all measurements recorded in the first 12 hours after dosing.
Time Frame: Baseline and Week 6.
Population: Full analysis set with last observation carried forward.
Measure: Least Squares Mean (Standard Error); unit: mmHg
Arm/Group | Azilsartan Medoxomil 20 mg QD | Azilsartan Medoxomil 40 mg QD | Azilsartan Medoxomil 80 mg QD | Olmesartan 40 mg QD | Placebo QD
Number analyzed (Participants) | 241 | 244 | 243 | 250 | 120
mmHg | -7.72 (0.519) | -8.63 (0.516) | -8.88 (0.517) | -7.86 (0.510) | -0.47 (0.736)
Statistical Analysis 1: Comparison: Azilsartan Medoxomil 20 mg QD vs Placebo QD; Test type: Superiority or Other; p < 0.001, ANCOVA — [p-value comment as in outcome 3, analysis 1]; Mean Difference (Final Values) = -7.25, 95% CI 2-sided [-9.02 to -5.48]
Statistical Analysis 2: Comparison: Azilsartan Medoxomil 40 mg QD vs Placebo QD; Test type: Superiority or Other; p < 0.001, ANCOVA — [p-value comment as in outcome 3, analysis 1]; Mean Difference (Final Values) = -8.16, 95% CI 2-sided [-9.92 to -6.40]
Statistical Analysis 3: Comparison: Azilsartan Medoxomil 80 mg QD vs Placebo QD; Test type: Superiority or Other; p < 0.001, ANCOVA — [p-value comment as in outcome 3, analysis 1]; Mean Difference (Final Values) = -8.41, 95% CI 2-sided [-10.17 to -6.65]
Statistical Analysis 4: Comparison: Azilsartan Medoxomil 20 mg QD vs Olmesartan 40 mg QD; Test type: Superiority or Other; p = 0.845, ANCOVA — [p-value comment as in outcome 3, analysis 1]; Mean Difference (Final Values) = 0.14, 95% CI 2-sided [-1.29 to 1.57]
Statistical Analysis 5: Comparison: Azilsartan Medoxomil 40 mg QD vs Olmesartan 40 mg QD; Test type: Superiority or Other; p = 0.290, ANCOVA — [p-value comment as in outcome 3, analysis 1]; Mean Difference (Final Values) = -0.77, 95% CI 2-sided [-2.19 to 0.65]
Statistical Analysis 6: Comparison: Azilsartan Medoxomil 80 mg QD vs Olmesartan 40 mg QD; Test type: Superiority or Other; p = 0.161, ANCOVA — [p-value comment as in outcome 3, analysis 1]; Mean Difference (Final Values) = -1.02, 95% CI 2-sided [-2.44 to 0.41]

11. Secondary Outcome: Change From Baseline in the Trough (22-24-hr) Mean Systolic Blood Pressure Measured by Ambulatory Blood Pressure Monitoring.
Description: The change in trough mean systolic blood pressure measured at week 6 relative to baseline. Ambulatory blood pressure monitoring measures blood pressure at regular intervals throughout the day and night. The trough mean is the average of all measurements recorded from 22 to 24 hours after dosing.
Time Frame: Baseline and Week 6.
Population: Full analysis set with last observation carried forward.
Measure: Least Squares Mean (Standard Error); unit: mmHg
Arm/Group | Azilsartan Medoxomil 20 mg QD | Azilsartan Medoxomil 40 mg QD | Azilsartan Medoxomil 80 mg QD | Olmesartan 40 mg QD | Placebo QD
Number analyzed (Participants) | 241 | 244 | 242 | 250 | 120
mmHg | -12.15 (0.864) | -12.39 (0.858) | -13.42 (0.862) | -11.10 (0.848) | -1.21 (1.224)
Statistical Analysis 1: Comparison: Azilsartan Medoxomil 20 mg QD vs Placebo QD; Test type: Superiority or Other; p < 0.001, ANCOVA — [p-value comment as in outcome 3, analysis 1]; Mean Difference (Final Values) = -10.94, 95% CI 2-sided [-13.88 to -8.00]
Statistical Analysis 2: Comparison: Azilsartan Medoxomil 40 mg QD vs Placebo QD; Test type: Superiority or Other; p < 0.001, ANCOVA — [p-value comment as in outcome 3, analysis 1]; Mean Difference (Final Values) = -11.18, 95% CI 2-sided [-14.11 to -8.24]
Statistical Analysis 3: Comparison: Azilsartan Medoxomil 80 mg QD vs Placebo QD; Test type: Superiority or Other; p < 0.001, ANCOVA — [p-value comment as in outcome 3, analysis 1]; Mean Difference (Final Values) = -12.21, 95% CI 2-sided [-15.15 to -9.28]
Statistical Analysis 4: Comparison: Azilsartan Medoxomil 20 mg QD vs Olmesartan 40 mg QD; Test type: Superiority or Other; p = 0.385, ANCOVA — [p-value comment as in outcome 3, analysis 1]; Mean Difference (Final Values) = -1.05, 95% CI 2-sided [-3.43 to 1.33]
Statistical Analysis 5: Comparison: Azilsartan Medoxomil 40 mg QD vs Olmesartan 40 mg QD; Test type: Superiority or Other; p = 0.285, ANCOVA — [p-value comment as in outcome 3, analysis 1]; Mean Difference (Final Values) = -1.29, 95% CI 2-sided [-3.66 to 1.08]
Statistical Analysis 6: Comparison: Azilsartan Medoxomil 80 mg QD vs Olmesartan 40 mg QD; Test type: Superiority or Other; p = 0.054, ANCOVA — [p-value comment as in outcome 3, analysis 1]; Mean Difference (Final Values) = -2.33, 95% CI 2-sided [-4.70 to 0.04]

12. Secondary Outcome: Change From Baseline in the Trough (22-24-hr) Mean Diastolic Blood Pressure Measured by Ambulatory Blood Pressure Monitoring.
Description: The change in trough mean diastolic blood pressure measured at week 6 relative to baseline. Ambulatory blood pressure monitoring measures blood pressure at regular intervals throughout the day and night. The trough mean is the average of all measurements recorded from 22 to 24 hours after dosing.
Time Frame: Baseline and Week 6.
Population: Full analysis set with last observation carried forward.
Measure: Least Squares Mean (Standard Error); unit: mmHg
Arm/Group | Azilsartan Medoxomil 20 mg QD | Azilsartan Medoxomil 40 mg QD | Azilsartan Medoxomil 80 mg QD | Olmesartan 40 mg QD | Placebo QD
Number analyzed (Participants) | 241 | 244 | 242 | 250 | 120
mmHg | -7.96 (0.614) | -7.93 (0.610) | -8.68 (0.612) | -7.56 (0.603) | -1.12 (0.870)
Statistical Analysis 1: Comparison: Azilsartan Medoxomil 20 mg QD vs Placebo QD; Test type: Superiority or Other; p < 0.001, ANCOVA — [p-value comment as in outcome 3, analysis 1]; Mean Difference (Final Values) = -6.84, 95% CI 2-sided [-8.93 to -4.75]
Statistical Analysis 2: Comparison: Azilsartan Medoxomil 40 mg QD vs Placebo QD; Test type: Superiority or Other; p < 0.001, ANCOVA — [p-value comment as in outcome 3, analysis 1]; Mean Difference (Final Values) = -6.80, 95% CI 2-sided [-8.89 to -4.72]
Statistical Analysis 3: Comparison: Azilsartan Medoxomil 80 mg QD vs Placebo QD; Test type: Superiority or Other; p < 0.001, ANCOVA — [p-value comment as in outcome 3, analysis 1]; Mean Difference (Final Values) = -7.55, 95% CI 2-sided [-9.64 to -5.47]
Statistical Analysis 4: Comparison: Azilsartan Medoxomil 20 mg QD vs Olmesartan 40 mg QD; Test type: Superiority or Other; p = 0.642, ANCOVA — [p-value comment as in outcome 3, analysis 1]; Mean Difference (Final Values) = -0.40, 95% CI 2-sided [-2.09 to 1.29]
Statistical Analysis 5: Comparison: Azilsartan Medoxomil 40 mg QD vs Olmesartan 40 mg QD; Test type: Superiority or Other; p = 0.672, ANCOVA — [p-value comment as in outcome 3, analysis 1]; Mean Difference (Final Values) = -0.36, 95% CI 2-sided [-2.05 to 1.32]
Statistical Analysis 6: Comparison: Azilsartan Medoxomil 80 mg QD vs Olmesartan 40 mg QD; Test type: Superiority or Other; p = 0.196, ANCOVA — [p-value comment as in outcome 3, analysis 1]; Mean Difference (Final Values) = -1.11, 95% CI 2-sided [-2.80 to 0.57]

13. Secondary Outcome: Percentage of Participants Who Achieve a Clinic Systolic Blood Pressure Response, Defined as < 140 mm Hg and/or Reduction From Baseline ≥ 20 mm Hg
Description: Percentage of participants who achieve a clinic systolic blood pressure response measured at week 6, defined as less than 140 mm Hg and/or reduction from baseline of greater than or equal to 20 mm Hg. Systolic blood pressure is the arithmetic mean of the 3 trough sitting systolic blood pressure measurements.
Time Frame: Baseline and Week 6.
Population: Full analysis set with last observation carried forward.
Measure: Number; unit: percentage of participants
Arm/Group | Azilsartan Medoxomil 20 mg QD | Azilsartan Medoxomil 40 mg QD | Azilsartan Medoxomil 80 mg QD | Olmesartan 40 mg QD | Placebo QD
Number analyzed (Participants) | 274 | 276 | 279 | 281 | 140
percentage of participants | 47.8 | 50.4 | 56.6 | 53.2 | 17.1
Statistical Analysis 1: Comparison: Azilsartan Medoxomil 20 mg QD vs Placebo QD; Test type: Superiority or Other; p < 0.001, Regression, Logistic — P-value for response criteria for systolic blood pressure was from a logistic regression with treatment as a factor and baseline clinic systolic blood pressure as a covariate. The unadjusted p-value is presented; Odds Ratio (OR) = 4.48, 95% CI 2-sided [2.71 to 7.39]
Statistical Analysis 2: Comparison: Azilsartan Medoxomil 40 mg QD vs Placebo QD; Test type: Superiority or Other; p < 0.001, Regression, Logistic — [p-value comment as in outcome 13, analysis 1]; Odds Ratio (OR) = 4.97, 95% CI 2-sided [3.01 to 8.20]
Statistical Analysis 3: Comparison: Azilsartan Medoxomil 80 mg QD vs Placebo QD; Test type: Superiority or Other; p < 0.001, Regression, Logistic — [p-value comment as in outcome 13, analysis 1]; Odds Ratio (OR) = 6.53, 95% CI 2-sided [3.95 to 10.79]
Statistical Analysis 4: Comparison: Azilsartan Medoxomil 20 mg QD vs Olmesartan 40 mg QD; Test type: Superiority or Other; p = 0.173, Regression, Logistic — [p-value comment as in outcome 13, analysis 1]; Odds Ratio (OR) = 0.79, 95% CI 2-sided [0.57 to 1.11]
Statistical Analysis 5: Comparison: Azilsartan Medoxomil 40 mg QD vs Olmesartan 40 mg QD; Test type: Superiority or Other; p = 0.449, Regression, Logistic — [p-value comment as in outcome 13, analysis 1]; Odds Ratio (OR) = 0.88, 95% CI 2-sided [0.63 to 1.23]
Statistical Analysis 6: Comparison: Azilsartan Medoxomil 80 mg QD vs Olmesartan 40 mg QD; Test type: Superiority or Other; p = 0.402, Regression, Logistic — [p-value comment as in outcome 13, analysis 1]; Odds Ratio (OR) = 1.15, 95% CI 2-sided [0.83 to 1.62]

14. Secondary Outcome: Percentage of Participants Who Achieve a Clinic Diastolic Blood Pressure Response, Defined as < 90 mm Hg and/or Reduction From Baseline ≥ 10 mm Hg
Description: Percentage of participants who achieve a clinic diastolic blood pressure response measured at week 6, defined as less than 90 mm Hg and/or reduction from baseline of greater than or equal to 10 mm Hg. Diastolic blood pressure is the arithmetic mean of the 3 trough sitting diastolic blood pressure measurements.
Time Frame: Baseline and Week 6.
Population: Full analysis set with last observation carried forward.
Measure: Number; unit: percentage of participants
Arm/Group | Azilsartan Medoxomil 20 mg QD | Azilsartan Medoxomil 40 mg QD | Azilsartan Medoxomil 80 mg QD | Olmesartan 40 mg QD | Placebo QD
Number analyzed (Participants) | 274 | 276 | 279 | 281 | 140
percentage of participants | 67.5 | 71.0 | 73.5 | 73.9 | 47.9
Statistical Analysis 1: Comparison: Azilsartan Medoxomil 20 mg QD vs Placebo QD; Test type: Superiority or Other; p < 0.001, Regression, Logistic — P-value for response criteria for diastolic blood pressure was from a logistic regression with treatment as a factor and baseline clinic diastolic blood pressure as a covariate. The unadjusted p-value is presented; Odds Ratio (OR) = 2.86, 95% CI 2-sided [1.82 to 4.48]
Statistical Analysis 2: Comparison: Azilsartan Medoxomil 40 mg QD vs Placebo QD; Test type: Superiority or Other; p < 0.001, Regression, Logistic — [p-value comment as in outcome 14, analysis 1]; Odds Ratio (OR) = 3.39, 95% CI 2-sided [2.15 to 5.35]
Statistical Analysis 3: Comparison: Azilsartan Medoxomil 80 mg QD vs Placebo QD; Test type: Superiority or Other; p < 0.001, Regression, Logistic — [p-value comment as in outcome 14, analysis 1]; Odds Ratio (OR) = 3.81, 95% CI 2-sided [2.41 to 6.02]
Statistical Analysis 4: Comparison: Azilsartan Medoxomil 20 mg QD vs Olmesartan 40 mg QD; Test type: Superiority or Other; p = 0.177, Regression, Logistic — [p-value comment as in outcome 14, analysis 1]; Odds Ratio (OR) = 0.76, 95% CI 2-sided [0.52 to 1.13]
Statistical Analysis 5: Comparison: Azilsartan Medoxomil 40 mg QD vs Olmesartan 40 mg QD; Test type: Superiority or Other; p = 0.628, Regression, Logistic — [p-value comment as in outcome 14, analysis 1]; Odds Ratio (OR) = 0.91, 95% CI 2-sided [0.61 to 1.35]
Statistical Analysis 6: Comparison: Azilsartan Medoxomil 80 mg QD vs Olmesartan 40 mg QD; Test type: Superiority or Other; p = 0.928, Regression, Logistic — [p-value comment as in outcome 14, analysis 1]; Odds Ratio (OR) = 1.02, 95% CI 2-sided [0.68 to 1.52]

15. Secondary Outcome: Percentage of Participants Who Achieve Both a Clinic Diastolic and Systolic Blood Pressure Response
Description: Percentage of participants who achieve both a clinic diastolic and systolic blood pressure response measured at week 6, defined as less than 90 mm Hg and/or reduction from baseline of greater than or equal to 10 mm Hg AND less than 140 mm Hg and/or reduction from baseline of greater than or equal to 20 mm Hg. Diastolic and systolic blood pressure is based on the arithmetic mean of the 3 sitting blood pressure measurements.
Time Frame: Baseline and Week 6.
Population: Full analysis set with last observation carried forward.
Measure: Number; unit: percentage of participants
Arm/Group | Azilsartan Medoxomil 20 mg QD | Azilsartan Medoxomil 40 mg QD | Azilsartan Medoxomil 80 mg QD | Olmesartan 40 mg QD | Placebo QD
Number analyzed (Participants) | 274 | 276 | 279 | 281 | 140
percentage of participants | 42.7 | 45.3 | 52.0 | 47.5 | 14.3
Statistical Analysis 1: Comparison: Azilsartan Medoxomil 20 mg QD vs Placebo QD; Test type: Superiority or Other; p < 0.001, Regression, Logistic — P-value for joint response criteria for systolic blood pressure and diastolic blood pressure was from a logistic regression with treatment as a factor and baseline clinic systolic blood pressure as a covariate. The unadjusted p-value is presented; Odds Ratio (OR) = 4.53, 95% CI 2-sided [2.66 to 7.72]
Statistical Analysis 2: Comparison: Azilsartan Medoxomil 40 mg QD vs Placebo QD; Test type: Superiority or Other; p < 0.001, Regression, Logistic — [p-value comment as in outcome 15, analysis 1]; Odds Ratio (OR) = 5.04, 95% CI 2-sided [2.96 to 8.58]
Statistical Analysis 3: Comparison: Azilsartan Medoxomil 80 mg QD vs Placebo QD; Test type: Superiority or Other; p < 0.001, Regression, Logistic — [p-value comment as in outcome 15, analysis 1]; Odds Ratio (OR) = 6.75, 95% CI 2-sided [3.96 to 11.48]
Statistical Analysis 4: Comparison: Azilsartan Medoxomil 20 mg QD vs Olmesartan 40 mg QD; Test type: Superiority or Other; p = 0.217, Regression, Logistic — [p-value comment as in outcome 15, analysis 1]; Odds Ratio (OR) = 0.81, 95% CI 2-sided [0.58 to 1.13]
Statistical Analysis 5: Comparison: Azilsartan Medoxomil 40 mg QD vs Olmesartan 40 mg QD; Test type: Superiority or Other; p = 0.537, Regression, Logistic — [p-value comment as in outcome 15, analysis 1]; Odds Ratio (OR) = 0.90, 95% CI 2-sided [0.64 to 1.26]
Statistical Analysis 6: Comparison: Azilsartan Medoxomil 80 mg QD vs Olmesartan 40 mg QD; Test type: Superiority or Other; p = 0.276, Regression, Logistic — [p-value comment as in outcome 15, analysis 1]; Odds Ratio (OR) = 1.20, 95% CI 2-sided [0.86 to 1.68]

ADVERSE EVENTS:
Time Frame: Treatment-emergent adverse events are adverse events that started after the first dose of double-blind study drug and no more than 14 days (or 30 days for a serious adverse event) after the last dose of double-blind study drug.
Description: At each visit the investigator had to document any occurrence of adverse events and abnormal laboratory findings. Any event spontaneously reported by the participant or observed by the investigator was recorded, irrespective of the relation to study treatment.
Arm/Group | Azilsartan Medoxomil 20 mg QD | Azilsartan Medoxomil 40 mg QD | Azilsartan Medoxomil 80 mg QD | Olmesartan 40 mg QD | Placebo QD
Serious Adverse Events (participants affected / at risk) | 8/283 | 0/281 | 1/284 | 2/282 | 3/142
Other Adverse Events (participants affected / at risk) | 23/283 | 19/281 | 32/284 | 18/282 | 13/142
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Azilsartan Medoxomil 20 mg QD (N=283) | Azilsartan Medoxomil 40 mg QD (N=281) | Azilsartan Medoxomil 80 mg QD (N=284) | Olmesartan 40 mg QD (N=282) | Placebo QD (N=142)
Atrial fibrillation (Cardiac disorders) | 1 | 0 | 0 | 0 | 0
Coronary artery disease (Cardiac disorders) | 0 | 0 | 0 | 0 | 1
Myocardial infarction (Cardiac disorders) | 1 | 0 | 0 | 0 | 0
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0
Inguinal hernia (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0
Chest pain (General disorders) | 0 | 0 | 0 | 0 | 1
Cholecystitis chronic (Hepatobiliary disorders) | 0 | 0 | 0 | 1 | 0
Cellulitis (Infections and infestations) | 1 | 0 | 0 | 0 | 0
Lower respiratory tract infection (Infections and infestations) | 1 | 0 | 0 | 0 | 0
Pneumonia (Infections and infestations) | 1 | 0 | 0 | 0 | 0
Myelodysplastic syndrome (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 0 | 0
Epilepsy (Nervous system disorders) | 1 | 0 | 0 | 0 | 0
Ischaemic stroke (Nervous system disorders) | 1 | 0 | 0 | 0 | 0
Transient ischaemic attack (Nervous system disorders) | 0 | 0 | 1 | 0 | 0
Status asthmaticus (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 | 0
Ischaemia (Vascular disorders) | 0 | 0 | 0 | 0 | 1
Shock (Vascular disorders) | 1 | 0 | 0 | 0 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Azilsartan Medoxomil 20 mg QD (N=283) | Azilsartan Medoxomil 40 mg QD (N=281) | Azilsartan Medoxomil 80 mg QD (N=284) | Olmesartan 40 mg QD (N=282) | Placebo QD (N=142)
Headache (Nervous system disorders) | 13 | 9 | 16 | 9 | 10
Dyslipidemia (Metabolism and nutrition disorders) | 10 | 11 | 16 | 10 | 3

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
No publication related to study results will be published prior to publication of a multi-center report submitted for publication within 18 months after conclusion or termination of a study at all study sites. Results publications will be submitted to sponsor for review 60 days in advance of publication. Sponsor can require removal of confidential information unrelated to study results. Sponsor can embargo a proposed publication for another 60 days to preserve intellectual property.